CLINICAL TRIAL: NCT04758910
Title: The Effect of High Flow Oxygen Therapy Via Tracheostomy on Diaphragm Function in Patients With Prolonged Weaning From Mechanical Ventilation
Brief Title: The Effect of High Flow Oxygen Therapy Via Tracheostomy on Diaphragm Function
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Evangelismos Hospital (Other)
Responsible Party: Principal Investigator, CHRISTINA ROUTSI, Professor in Medicine, National and Kapodistrian University of Athens, Athens, Greece, Evangelismos Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: No 771 2019
Record Dates: First submitted 2021-01-19; First posted 2021-02-17 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Weaning Failure
Keywords: prolonged weaning; tracheostomy; high flow oxygen therapy

STUDY DESIGN:
Intervention Model Description: Participants will receive two treatments : high flow oxygen therapy and T-piece.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Flow Oxygen Therapy (Active Comparator): Tracheostomized patients will undergo a spontaneous breathing trial with high flow oxygen therapy.
  Interventions: Device: High Flow Oxygen Therapy
- T-piece (Active Comparator): Tracheostomized patients will undergo a spontaneous breathing trial with T-piece as a standard of care.
  Interventions: Device: T-piece

INTERVENTIONS:
Device: High Flow Oxygen Therapy — A 30-minute spontaneous breathing trial using high flow oxygen therapy via tracheostomy.
  Arms: High Flow Oxygen Therapy
Device: T-piece — A 30-minute spontaneous breathing trial using T-piece via tracheostomy.
  Other Names: Standard of care
  Arms: T-piece

SUMMARY:
While the high flow oxygen therapy (HFOT) respiratory support system, delivered through nasal cannulas, has demonstrated clinical benefits on respiratory function, limited data exist on whether such effects are also present in HFOT through tracheostomy. Therefore, the aim of the proposed study is to examine the short-term effects of HFOT as opposed to oxygen therapy via T-piece on diaphragmatic function in tracheostomized patients with prolonged weaning from mechanical ventilation.

DETAILED DESCRIPTION:
Critically ill patients who experience difficulties in weaning from the ventilator often undergo tracheostomy. These patients usually undergo spontaneous breathing trials receiving oxygen via T-piece. While the high flow oxygen therapy (HFOT) respiratory support system, delivered through nasal cannulas, has demonstrated clinical benefits on respiratory function, limited data exist on whether such effects are also present in HFOT through tracheostomy. Therefore, we plan to perform a study to examine the short-term effects of HFOT on diaphragmatic function in tracheostomized patients with prolonged weaning from mechanical ventilation.

After disconnection from the ventilator, patients will undergo a 30-minute spontaneous breathing trial receiving oxygen either conventionally via T-piece, or by HFOT delivered via tracheostomy, followed by a washout period of 15 min breathing through T-piece and 30 min receiving oxygen with the other modality in a randomized manner. At the start and end of each study period, patients will undergo an assessment through diaphragm ultrasonography, which includes excursion of diaphragmatic dome and thickness of diaphragmatic zone of apposition at end-inspiration and end-expiration. Subsequently, the diaphragmatic thickening fraction will be calculated as the difference between end-inspiratory and end-expiratory thickness divided by end-expiratory thickness. Also. arterial blood gases as well as respiratory rate (RR) and tidal volume (TV) (through a Wright's spirometer) will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Mechanically ventilated patients with prolonged weaning and tracheostomy

Exclusion Criteria:

* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-03-01 (Estimated); Primary Completion 2021-05-30 (Estimated); Study Completion 2021-07-30 (Estimated)

PRIMARY OUTCOMES:
Diaphragmatic function | 30 minutes
  Differences in diaphragmatic function between high flow oxygen therapy and T-piece will be assessed by diaphragm excursion measurement (in cm) using bedside ultrasound examination of the diaphragm.
Diaphragmatic thickening fraction | 30 minutes
  Differences in diaphragmatic thickening fraction between high flow oxygen therapy and T-piece will be assessed using bedside ultrasound examination of the diaphragm thickness of diaphragmatic zone of apposition at end-inspiration and end-expiration and subsequent calculation of the difference between end-inspiratory and end-expiratory thickness divided by end-expiratory thickness.

SECONDARY OUTCOMES:
Tidal volume | 30 minutes
  Differences in tidal volume between high flow oxygen therapy and T-piece will be assessed by tidal volume (in mL) measurement by a Wright's spirometer.
Respiratory frequence | 30 minutes
  Differences in respiratory frequency between high flow oxygen therapy and T-piece will be assessed by respiratory rate measurement (breaths per minute).

REFERENCES:
- [Background] Beduneau G, Pham T, Schortgen F, Piquilloud L, Zogheib E, Jonas M, Grelon F, Runge I, Nicolas Terzi, Grange S, Barberet G, Guitard PG, Frat JP, Constan A, Chretien JM, Mancebo J, Mercat A, Richard JM, Brochard L; WIND (Weaning according to a New Definition) Study Group and the REVA (Reseau Europeen de Recherche en Ventilation Artificielle) Network double dagger. Epidemiology of Weaning Outcome according to a New Definition. The WIND Study. Am J Respir Crit Care Med. 2017 Mar 15;195(6):772-783. doi: 10.1164/rccm.201602-0320OC. PMID 27626706
- [Background] Kim WY, Suh HJ, Hong SB, Koh Y, Lim CM. Diaphragm dysfunction assessed by ultrasonography: influence on weaning from mechanical ventilation. Crit Care Med. 2011 Dec;39(12):2627-30. doi: 10.1097/CCM.0b013e3182266408. PMID 21705883
- [Background] Matamis D, Soilemezi E, Tsagourias M, Akoumianaki E, Dimassi S, Boroli F, Richard JC, Brochard L. Sonographic evaluation of the diaphragm in critically ill patients. Technique and clinical applications. Intensive Care Med. 2013 May;39(5):801-10. doi: 10.1007/s00134-013-2823-1. Epub 2013 Jan 24. PMID 23344830
- [Background] Frat JP, Thille AW, Mercat A, Girault C, Ragot S, Perbet S, Prat G, Boulain T, Morawiec E, Cottereau A, Devaquet J, Nseir S, Razazi K, Mira JP, Argaud L, Chakarian JC, Ricard JD, Wittebole X, Chevalier S, Herbland A, Fartoukh M, Constantin JM, Tonnelier JM, Pierrot M, Mathonnet A, Beduneau G, Deletage-Metreau C, Richard JC, Brochard L, Robert R; FLORALI Study Group; REVA Network. High-flow oxygen through nasal cannula in acute hypoxemic respiratory failure. N Engl J Med. 2015 Jun 4;372(23):2185-96. doi: 10.1056/NEJMoa1503326. Epub 2015 May 17. PMID 25981908
- [Background] Stripoli T, Spadaro S, Di Mussi R, Volta CA, Trerotoli P, De Carlo F, Iannuzziello R, Sechi F, Pierucci P, Staffieri F, Bruno F, Camporota L, Grasso S. High-flow oxygen therapy in tracheostomized patients at high risk of weaning failure. Ann Intensive Care. 2019 Jan 7;9(1):4. doi: 10.1186/s13613-019-0482-2. PMID 30617626
- [Background] Natalini D, Grieco DL, Santantonio MT, Mincione L, Toni F, Anzellotti GM, Eleuteri D, Di Giannatale P, Antonelli M, Maggiore SM. Physiological effects of high-flow oxygen in tracheostomized patients. Ann Intensive Care. 2019 Oct 7;9(1):114. doi: 10.1186/s13613-019-0591-y. PMID 31591659
- [Background] Delorme M, Bouchard PA, Simon M, Simard S, Lellouche F. Effects of High-Flow Nasal Cannula on the Work of Breathing in Patients Recovering From Acute Respiratory Failure. Crit Care Med. 2017 Dec;45(12):1981-1988. doi: 10.1097/CCM.0000000000002693. PMID 28857852
- [Derived] Lytra E, Kokkoris S, Poularas I, Filippiadis D, Cokkinos D, Exarhos D, Zakynthinos S, Routsi C. The effect of high-flow oxygen via tracheostomy on respiratory pattern and diaphragmatic function in patients with prolonged mechanical ventilation: A randomized, physiological, crossover study. J Intensive Med. 2024 Jan 4;4(2):202-208. doi: 10.1016/j.jointm.2023.11.008. eCollection 2024 Apr. PMID 38681788